CLINICAL TRIAL: NCT00370084
Title: Effects of Itopride Hydrochloride on Gastric Emptying, Glycaemia and "Meal-related" Symptoms in Patients With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Itopride Hydrochloride in Diabetes: Effects on Gastric Emptying and Glycemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITODG04-01; 041026
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — itopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Itopride (Experimental)
  Interventions: Drug: Itopride

INTERVENTIONS:
Drug: Itopride — oral, three times daily
  Arms: Itopride
Other: Placebo — oral, three times daily
  Arms: Placebo

SUMMARY:
Itopride is a new compound that is already marketed in Japan and in some countries of Eastern Europe under the name of Ganaton. It is used to treat symptoms associated with gastroparesis. Due to inadequate gastric emptying, these patients often have symptoms of bloating, nausea and vomiting following ingestion of a meal. The goal of this study is to evaluate the effects of Itopride on gastric motor function and glycemia in patients with diabetes.

DETAILED DESCRIPTION:
This is a mechanistic study evaluating in a cross-over design the effects of Itopride hydrochloride.

The primary objective of this study is to evaluate the acute effects of itopride hydrochloride (200 mg three times daily) on gastric emptying of solid and liquid meal components in patients with type 1 and type 2 diabetes mellitus. Secondary objectives are to evaluate the effects of itopride hydrochloride on the glycaemic response to a meal, "meal-related" upper gastrointestinal symptoms and intragastric meal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Type-1 and Type-2 diabetic patients
* 18 to 65 years old
* Glycated haemoglobin level (HbA1c) below 9%
* Body mass index (BMI) between 18 and 35 kg/m2

Exclusion Criteria:

* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study (e.g. prokinetic drugs, macrolide antibiotics)
* Exposure to radiation for research purposes during the previous 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Gastric emptying assessment | weekly

SECONDARY OUTCOMES:
Glycemia, relief of upper gastrointestinal symptoms, intragastric meal distribution | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Michael Horowitz, M.D., Principal Investigator — Royal Adelaide Hospital
Locations (1):
- University of Adelaide, Department of Medicine, Adelaide, South Australia, Australia